

taking consent







Version 2 20-Feb-19 Centre: PIN: REC Number: IRAS ID: 256260

## PARTICIPANT CONSENT FORM FOR PARENTS/CARERS

## This consent form is for parents/carers who wish to take part in the study

## Online PTSD treatment for Young People and their Carers (OPTYC): Case Series Dr Patrick Smith

| | ve had the opportunity to o | neet dated13/12/18 (version 1.0) for the consider the information, ask questions and have |
|---|---|---|
| 2. I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. | | |
| <ol> <li>I understand that the information collected about me will be used to support other research in the future, and may be shared anonymously with other researchers.</li> <li>I understand that the information held and maintained by South London and Maudsley NHS Foundation Trust may be used to help contact me or provide information about my health status.</li> </ol> | | |
| 6. I agree to take pa | art in the above study. | |
| lame of Participant | Date | Signature |
| lame of Person | <br>Date | Signature |